CLINICAL TRIAL: NCT06105840
Title: Effect of Combination of Curcuminoid Standardized Turmeric Extract With Acupressure on Inflammatory Markers, Endorphins and Quality of Life in Elderly People With Osteoarthritis Genu
Brief Title: Combination of Curcuminoid With Acupressure for Inflammation and Pain in the Elderly With Osteoarthritis Genu
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Srinalesti Mahanani, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KE/FK/0674/EC/2023
Record Dates: First submitted 2023-10-02; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
Keywords: curcuminoid; acupressure; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Groups assigned randomly using lottery draw number 1
  Interventions: Procedure: Acupressure and Standardized Curcuminoid from Turmeric Extract
- Control Group (Sham Comparator): Groups assigned randomly using lottery draw number 2
  Interventions: Procedure: Sham Acupressure and Placebo

INTERVENTIONS:
Procedure: Acupressure and Standardized Curcuminoid from Turmeric Extract — capsules containing curcuminoid from Tumeric Extract three times a day for 3 weeks and acupressure massage at points provide comfort for knee pain twice a week for 3 weeks
  Arms: Intervention Group
Procedure: Sham Acupressure and Placebo — capsules containing starch three times a day for 3 weeks and acupressure massage at points that are not to provide comfort for knee pain twice a week for 3 weeks
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to to investigate the efficacy of acupressure and standardized curcuminoids from turmeric extract to inflammatory markers, endorphin hormones in the blood and quality of life in elderly patient with Osteoarthritis Genu.

The main questions it aims to answer are:

1. Is there any effect combination of acupressure and standardized curcuminoids from turmeric extract to inflammatory markers in elderly patients with Osteoarthritis Genu?
2. Is there any effect combination of acupressure and standardized curcuminoids from turmeric extract to endorphin hormones in the blood in elderly patients with Osteoarthritis Genu?
3. Is there an effect combination of acupressure and standardized curcuminoids from turmeric extract to quality of life in elderly patients with Osteoarthritis Genu?

Participants in the intervention group received 2 treatments, namely acupressure at points that provide osteoarthritis-specific comfort and standardized curcuminoids from turmeric extract capsules. Participant in the control group alo would receive 2 treatments, an active placebo (starch capsules and sham acupressure).

Researchers will compare interventional group and sham group to see efficacy the combination therapy

DETAILED DESCRIPTION:
Background. One of the degeneration processes that occurs in the elderly is the musculoskeletal system. These deteriorations include bone loss and a decrease in joint fluid volume which is exacerbated by bearing the weight of the body. Pain in Osteoarthritis patients affects many areas of quality of life such as physical function, emotional behavior, and mental health. Osteoarthritis-related pain is a major factor in poor quality of life. The most common pharmacological treatment to control pain is the use of non-steroidal anti-inflammatory drugs (NSAIDs), but these drugs carry the risk of causing side effects. Limitations associated with pharmacologic treatment result in patients choosing commonly available alternative therapies for pain management. Popular alternative therapies include herbal therapy, therapeutic touch, relaxation techniques, music therapy, acupuncture, and acupressure. This alternative therapy, unlike the use of drugs, does not produce dangerous side effects.

Research on the effectiveness of herbal therapy on inflammatory osteoarthritis patients was conducted in Indonesia in 2009 on 80 sufferers with the result that administration of turmeric rhizome extract curcuminoids significantly suppressed the activity of synovial fluid monocytes to secrete Cyclooxygenase-2 (COX-2) and Reactive Oxygen Intermediate (ROI), reduced leukocyte numbers and fluid Malondialdehyde (MDA) levels. synovia and reduces Osteoarthritis (OA) joint pain, with an ability that is not significantly different compared to diclofenac sodium therapy 3x25 mg per day. Furthermore, the development of herbal therapy for Osteoathritis continued with research which proved that the combination of ginger, ginger, soybean and shrimp shell extracts provided significant results in reducing joint pain, stiffness and physical disability which were evaluated based on the Western Ontario and McMaster values. Universities Osteoarthritis Index (WOMAC) and did not show a significant difference when compared with meloxicam.

Research that has been carried out to evaluate the effectiveness of acupressure therapy for the pain of Osteoarthritis patients was also carried out in several countries, including by study on 40 Osteoarthritis patients who were divided into two groups (intervention and control). In the intervention group, acupressure therapy was given for 5 days with a duration of 30 minutes each time. The results showed that the average pain score in the intervention group decreased significantly from 5.89 at the beginning of the study to 4.11 at the end of the study, while the pain score did not change substantially in the control group. These findings remained consistent after adjusting for age, weight, and pretreatment covariates. This study supports the evidence that Acupressure therapy provides an effective option for short-term knee pain relief in patients with knee Osteoarthritis. In line with the results, there was research which was conducted on 51 elderly with osteoarthritis divided into 3 groups (acupressure intervention, placebo and control). This study revealed that respondents who received acupressure therapy for 3-4 weeks with the duration of each therapy being 10-15 minutes, showed a significant reduction in the total WOMAC index, pain and physical dysfunction.

So far, there has been no research combining standardized curcuminoid turmeric extract therapy with acupressure for inflammation and pain in osteoarthritis patients. More clinical trials with appropriate methodology are needed to confirm the effectiveness of standardized turmeric extract, curcuminoids and acupressure to treat physical problems in osteoarthritis patients.

Study Design/Methods. The research will be carried out by design Randomized Controlled Trials (RCT). Respondents will be divided randomly into 2 groups, namely treatment and control. The treatment group will receive interventions, namely herbal therapy and acupressure therapy, while the control group will receive active placebo (capsules containing starch and acupressure massage at points that are not to provide comfort for knee pain). In this study, a double blind technique was used , that is, the subjects and researchers did not know which respondents were in the treatment group and which respondents were in the control group.

Data Analysis Plan

1. Analysis Descriptive Data obtained done tabulation in accordance with general data grouping and special data results measurement variable pre-test and post-test research . Data analysis will used For get description general from each variable . Data processing uses distribution frequency , reading data distribution (mean, mode, median, etc deviation )
2. Analysis Inferential For know difference effectiveness on second group , researcher use Test the Difference with using the Independent T-Test and Wilcoxon Sign Rank Test. Analysis done on difference all over variable before And after done intervention on second group

ELIGIBILITY:
The inclusion criteria in this study are:

1. Clinical diagnosis of osteoarthritis which confirmed by physical examination and x-rays
2. Experience pain with a Numeric Rating scale of 1-7
3. Must be able to swallow capsules
4. Must be able to carry out mobility without assistance or with minimal assistance

The exclusion criteria in this study are:

1. Parkinson's disease
2. Dementia disease
3. Psychosis disease
4. New bone fractures
5. Joint dislocations
6. Cancer
7. Rheumatic diseases other than osteoarthritis (rheumatoid arthritis)
8. Undergoing joint replacement therapy.
9. Analgesic dependent disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-27 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Inflammation Marker | Outcome measurements will be carried out before starting therapy and after 3 weeks of therapy
  Inflammation markers are carried out by measuring Leukocyte Number, NLR, Blood Sediment Rate and COX-2 hormone. Outcome measurements will be carried out a complete blood test using a Hematology Analyzer. Leukocyte numbers measured in microliter (mcL). Neutrophil-Lymphocyte Count Ratio can be calculated from the number of neutrophils (cells) and lymphocytes (cells). Neutrophils and lymphocytes will be combined to report Neutrophil-Lymphocyte Count Ratio in %. Blood Sediment Rate is a measurement of the difference in the decrease in height of red blood cells in a test tube (mm) divided by the time (hours) required for all of them to settle to the bottom of the test tube. There will be combined to report Blood Sediment Rate in mm/hr. The COX-2 hormone examination was carried out using the Enzyme Linked Immunosorbent Assay (ELISA). The amount of COX-2 Hormone in the blood in nanograms and blood sample volume in milliliters will be combined to report secretion of COX-2 in ng/mL
Endorphin Hormones | Outcome measurements will be carried out before starting therapy and after 3 weeks of therapy
  Secretion of endorphin hormones Endorphins, in this case beta endorphin, are hormones released by the pituitary gland in response to stress or pain, which are also secreted in blood plasma. Endorphin hormone examination is carried out using the Enzyme Linked Immunosorbent Assay (ELISA) method on blood plasma. The amount of Endorphin Hormone in the blood in nanograms and the blood sample volume in milliliters will be combined to report secretion of COX-2 in ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Srinalesti Mahanani, Magister, Principal Investigator — Faculty of Medicine University of Gadjah Mada
Locations (1):
- Padukuhan Tanjungsari Kelurahan Sukoharjo Ngaglik, Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alinaghizadeh M, Hawkins J, Abbassian A, Seif Barghi T, Ayati MH, Alizadeh Vaghasloo M. Effect of Persian acupressure (Ghamz) on Patients with Knee Osteoarthritis: A Single-Blinded Parallel Clinical Trial. Pain Manag Nurs. 2021 Dec;22(6):820-827. doi: 10.1016/j.pmn.2021.06.002. Epub 2021 Jul 11. PMID 34261600
- [Result] Cheung DST, Yeung WF, Suen LK, Chong TC, Ho YS, Yu BY, Chan LY, Chen HY, Lao LX. Self-administered acupressure for knee osteoarthritis in middle-aged and older adults: a pilot randomized controlled trial. Acupunct Med. 2020 Apr;38(2):75-85. doi: 10.1177/0964528419883269. Epub 2019 Nov 13. PMID 31718229
- [Result] Guo D, Ma S, Zhao Y, Dong J, Guo B, Li X. Self-administered acupressure and exercise for patients with osteoarthritis: A randomized controlled trial. Clin Rehabil. 2022 Mar;36(3):350-358. doi: 10.1177/02692155211049155. Epub 2021 Oct 18. PMID 34658285
- [Result] Ho KK, Kwok AW, Chau WW, Xia SM, Wang YL, Cheng JC. A randomized controlled trial on the effect of focal thermal therapy at acupressure points treating osteoarthritis of the knee. J Orthop Surg Res. 2021 Apr 27;16(1):282. doi: 10.1186/s13018-021-02398-2. PMID 33906695
- [Result] Lee WJ, Park H. Effects of auricular acupressure on sleep and pain in elderly people who have osteoarthritis and live in nursing homes: A randomized, single-blind, placebo-controlled trial. Explore (NY). 2023 Mar-Apr;19(2):214-222. doi: 10.1016/j.explore.2022.07.001. Epub 2022 Jul 5. PMID 35835645
- [Result] Li LW, Harris RE, Tsodikov A, Struble L, Murphy SL. Self-Acupressure for Older Adults With Symptomatic Knee Osteoarthritis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Feb;70(2):221-229. doi: 10.1002/acr.23262. Epub 2017 Dec 29. PMID 28437570
- [Result] Sorour AS, Ayoub AS, Abd El Aziz EM. Effectiveness of acupressure versus isometric exercise on pain, stiffness, and physical function in knee osteoarthritis female patients. J Adv Res. 2014 Mar;5(2):193-200. doi: 10.1016/j.jare.2013.02.003. Epub 2013 Apr 8. PMID 25685487
- [Result] Kertia N, Asdie AH, Rochmah W, Marsetyawan. Ability of curcuminoid compared to diclofenac sodium in reducing the secretion of cycloxygenase-2 enzyme by synovial fluid's monocytes of patients with osteoarthritis. Acta Med Indones. 2012 Apr;44(2):105-13. PMID 22745140
- [Result] Adamczak A, Ozarowski M, Karpinski TM. Curcumin, a Natural Antimicrobial Agent with Strain-Specific Activity. Pharmaceuticals (Basel). 2020 Jul 16;13(7):153. doi: 10.3390/ph13070153. PMID 32708619
- [Result] Gomes TPO, Souza JIN, Somerlate LC, Mendonca VA, Lima NM, Carli GP, Castro SBR, de Jesus A S Andrade T, Dias JVL, Oliveira MAL, Alves CCS, Carli AP. Miconia albicans and Curcuma longa herbal medicines positively modulate joint pain, function and inflammation in patients with osteoarthritis: a clinical study. Inflammopharmacology. 2021 Apr;29(2):377-391. doi: 10.1007/s10787-020-00781-9. Epub 2021 Jan 16. PMID 33452967
- [Result] Kare SK, Vinay V, Maresz K, Prisk V, Vik H. Tamarindus indica Seed Extract-Based Botanical Compositions Alleviate Knee Pain and Improve Joint Function in Mild-to-Moderate Osteoarthritis: A Randomized, Double-Blind, Placebo-Controlled Clinical Study. Evid Based Complement Alternat Med. 2022 Jan 19;2022:2226139. doi: 10.1155/2022/2226139. eCollection 2022. PMID 35096104
- [Result] Madhu K, Chanda K, Saji MJ. Safety and efficacy of Curcuma longa extract in the treatment of painful knee osteoarthritis: a randomized placebo-controlled trial. Inflammopharmacology. 2013 Apr;21(2):129-36. doi: 10.1007/s10787-012-0163-3. Epub 2012 Dec 16. PMID 23242572
- [Result] Pinsornsak P, Niempoog S. The efficacy of Curcuma Longa L. extract as an adjuvant therapy in primary knee osteoarthritis: a randomized control trial. J Med Assoc Thai. 2012 Jan;95 Suppl 1:S51-8. PMID 23964444
- [Result] Rahimnia AR, Panahi Y, Alishiri G, Sharafi M, Sahebkar A. Impact of Supplementation with Curcuminoids on Systemic Inflammation in Patients with Knee Osteoarthritis: Findings from a Randomized Double-Blind Placebo-Controlled Trial. Drug Res (Stuttg). 2015 Oct;65(10):521-5. doi: 10.1055/s-0034-1384536. Epub 2014 Jul 22. PMID 25050518
- [Result] Raj JP, Venkatachalam S, Racha P, Bhaskaran S, Amaravati RS. Effect of Turmacin supplementation on joint discomfort and functional outcome among healthy participants - A randomized placebo-controlled trial. Complement Ther Med. 2020 Sep;53:102522. doi: 10.1016/j.ctim.2020.102522. Epub 2020 Jul 22. PMID 33066856
- [Result] Srivastava S, Saksena AK, Khattri S, Kumar S, Dagur RS. Curcuma longa extract reduces inflammatory and oxidative stress biomarkers in osteoarthritis of knee: a four-month, double-blind, randomized, placebo-controlled trial. Inflammopharmacology. 2016 Dec;24(6):377-388. doi: 10.1007/s10787-016-0289-9. Epub 2016 Oct 19. PMID 27761693
- [Result] Wan Y, Sun W, Yang J, Ren J, Kou Q. The comparison of curcuminoid formulations or its combination with conventional therapies versus conventional therapies alone for knee osteoarthritis. Clin Rheumatol. 2022 Jul;41(7):2153-2169. doi: 10.1007/s10067-022-06105-2. Epub 2022 Mar 16. PMID 35294665
- [Derived] Mahanani S, Kertia N, Madyaningrum E. Combination of Curcuminoids and Acupressure for Inflammation and Pain in Older People with Osteoarthritis Genu: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Jun 24;13:e54970. doi: 10.2196/54970. PMID 38771152
- See also: The effect of acupressure therapy on pain, stiffness and physical functioning of knees among older adults diagnosed with osteoarthritis: A pilot randomized control trial. — https://doi.org/10.1016/j.eujim.2019.04.007
- See also: Effectiveness of knee acupressure along with herbal knee poultice for knee osteoarthritis treatment: A pilot pre-post clinical study. — https://doi.org/10.1016/j.hermed.2021.100498
- See also: Effects of auricular acupressure on joint pain, range of motion, and sleep in the elderly with knee osteoarthritis — https://doi.org/10.12799/jkachn.2019.30.1.79
- See also: Adjunctive effects of acupressure therapy on pain and quality of life in patients with knee osteoarthritis: an interventional study. — https://doi.org/10.1007/s11726-021-1252-x
- See also: Acujoint, a highly efficient formulation with natural bioactive compounds, exerts potent anti-arthritis effects in human osteoarthritis - A pilot randomized double blind clinical study compared to combination of glucosamine and chondroitin — https://doi.org/10.1016/j.hermed.2019.100276

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT06105840/Prot_SAP_ICF_000.pdf